CLINICAL TRIAL: NCT03827915
Title: Double Sequence External Defibrillation: A Randomized Controlled Trial in Patients With Atrial Fibrillation Refractory to DC Cardioversion
Brief Title: Double Sequential External Defibrillation in Patients With Atrial Fibrillation Refractory to DC Cardioversion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2017-0457
Record Dates: First submitted 2019-01-28; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation; Defibrillators; Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Refractory atrial fibrillation; Double sequential external defibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Phase III, randomized controlled, superiority trial, with two parallel groups, conducted in one academic medical center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Third trial of DC cardioversion (No Intervention): Patients with atrial fibrillation who fail to revert to sinus rhythm after two failed DC cardioversion attempts will receive a third trial of DC cardioversion (Standard of care)
- Double sequential external defibrillation (Experimental): Patients with atrial fibrillation who fail to revert to sinus rhythm after two failed DC cardioversion attempts will receive DSED
  Interventions: Device: Double sequential external defibrillation

INTERVENTIONS:
Device: Double sequential external defibrillation — DSED is the process of using two defibrillators near simultaneously at their highest allowed energy setting and aims to treat refractory atrial fibrillation. The first set of pads is placed in the traditional anterolateral position and the second set can be either placed adjacent to the first set (antero-lateral) or in the antero-posterior position. Shocks are then delivered simultaneously or near simultaneously
  Arms: Double sequential external defibrillation

SUMMARY:
Atrial fibrillation (AF) is a common cardiac arrhythmia that leads to increased risk of heart failure, hospitalization, thromboembolic events, and death. Restoration of normal heart rhythm is performed in many patients with AF to improve symptoms. In this study, the investigators will consider patients who fail 2 or more trials of DC cardioversion as having refractory AF.

The aim of this study is to assess whether the use of double sequential defibrillation in patients with refractory AF has a higher success rate in reverting them to a normal heart rhythm than a third cardioversion.

This is a phase III, randomized controlled, single-centered, superiority trial. All patients with AF admitted to the coronary care unit (CCU) for DC cardioversion, and refractory to at least two trials of DC cardioversion will be enrolled. Patients are randomized into two arms: the first will receive a third trial of DC cardioversion (standard of care) and the second will receive double sequential external defibrillation.

The resolution of AF by reverting back to normal sinus rhythm is the primary outcome of the investigators. This will be determined using EKG (electrocardiogram) immediately after DC cardioversion or double sequential defibrillation.

DETAILED DESCRIPTION:
Patients presenting to the CCU with persistent AF for direct current (DC) cardioversion, who meet the inclusion criteria and fail to revert to normal sinus rhythm after two DC cardioversion attempts will be invited for enrollment in the study. No sampling will be carried out for the sake of this study.

Patients meeting the eligibility criteria will receive double sequential external defibrillation (DSED) or a third DC cardioversion (standard of care).

DSED is the process of using two defibrillators near simultaneously at their highest allowed energy setting and aims to treat refractory atrial fibrillation. The first set of pads is placed in the traditional anterolateral position and the second set can be either placed adjacent to the first set (antero-lateral) or in the antero-posterior position. Shocks are then delivered simultaneously or near simultaneously.

ELIGIBILITY:
Inclusion Criteria:

- Atrial Fibrillation patients admitted to the CCU for DC cardioversion, and refractory to at least two trials of DC cardioversion

Exclusion Criteria:

* Patients with Atrial Fibrillation not requiring DC cardioversion
* Patients with Atrial Fibrillation who reverted after a maximum of two trials of DC cardioversion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2024-01-21 (Estimated); Study Completion 2024-01-21 (Estimated)

PRIMARY OUTCOMES:
Number of participants with atrial fibrillation who revert back to normal sinus rhythm using Double Sequential External Defibrillation after two failed attempts of DC cardioversion. | 15 minutes
  Number of participants with atrial fibrillation who revert back to normal sinus rhythm using Double Sequential External Defibrillation after two failed attempts of DC cardioversion . This will be determined using an EKG (Electrocardiogram) immediately after double sequential external defibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Abou Dagher, M.D., Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Wolf PA, D'Agostino RB, Silbershatz H, Kannel WB, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. Circulation. 1998 Sep 8;98(10):946-52. doi: 10.1161/01.cir.98.10.946. PMID 9737513
- [Background] Chugh SS, Blackshear JL, Shen WK, Hammill SC, Gersh BJ. Epidemiology and natural history of atrial fibrillation: clinical implications. J Am Coll Cardiol. 2001 Feb;37(2):371-8. doi: 10.1016/s0735-1097(00)01107-4. PMID 11216949
- [Background] Patel NJ, Deshmukh A, Pant S, Singh V, Patel N, Arora S, Shah N, Chothani A, Savani GT, Mehta K, Parikh V, Rathod A, Badheka AO, Lafferty J, Kowalski M, Mehta JL, Mitrani RD, Viles-Gonzalez JF, Paydak H. Contemporary trends of hospitalization for atrial fibrillation in the United States, 2000 through 2010: implications for healthcare planning. Circulation. 2014 Jun 10;129(23):2371-9. doi: 10.1161/CIRCULATIONAHA.114.008201. Epub 2014 May 19. PMID 24842943
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Mead GE, Elder AT, Flapan AD, Kelman A. Electrical cardioversion for atrial fibrillation and flutter. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD002903. doi: 10.1002/14651858.CD002903.pub2. PMID 16034878
- [Background] Alam M, Thorstrand C. Left ventricular function in patients with atrial fibrillation before and after cardioversion. Am J Cardiol. 1992 Mar 1;69(6):694-6. doi: 10.1016/0002-9149(92)90169-y. No abstract available. PMID 1536123
- [Background] Xiong C, Sonnhag C, Nylander E, Wranne B. Atrial and ventricular function after cardioversion of atrial fibrillation. Br Heart J. 1995 Sep;74(3):254-60. doi: 10.1136/hrt.74.3.254. PMID 7547019
- [Background] Van Gelder IC, Crijns HJ, Blanksma PK, Landsman ML, Posma JL, Van Den Berg MP, Meijler FL, Lie KI. Time course of hemodynamic changes and improvement of exercise tolerance after cardioversion of chronic atrial fibrillation unassociated with cardiac valve disease. Am J Cardiol. 1993 Sep 1;72(7):560-6. doi: 10.1016/0002-9149(93)90352-d. PMID 8362771
- [Background] Jaakkola S, Lip GY, Biancari F, Nuotio I, Hartikainen JE, Ylitalo A, Airaksinen KE. Predicting Unsuccessful Electrical Cardioversion for Acute Atrial Fibrillation (from the AF-CVS Score). Am J Cardiol. 2017 Mar 1;119(5):749-752. doi: 10.1016/j.amjcard.2016.11.026. Epub 2016 Dec 2. PMID 28017305
- [Background] Levy S, Lauribe P, Dolla E, Kou W, Kadish A, Calkins H, Pagannelli F, Moyal C, Bremondy M, Schork A, et al. A randomized comparison of external and internal cardioversion of chronic atrial fibrillation. Circulation. 1992 Nov;86(5):1415-20. doi: 10.1161/01.cir.86.5.1415. PMID 1423954
- [Background] Kabukcu M, Demircioglu F, Yanik E, Minareci K, Ersel-Tuzuner F. Simultaneous double external DC shock technique for refractory atrial fibrillation in concomitant heart disease. Jpn Heart J. 2004 Nov;45(6):929-36. doi: 10.1536/jhj.45.929. PMID 15655268
- [Background] Chang MS, Inoue H, Kallok MJ, Zipes DP. Double and triple sequential shocks reduce ventricular defibrillation threshold in dogs with and without myocardial infarction. J Am Coll Cardiol. 1986 Dec;8(6):1393-405. doi: 10.1016/s0735-1097(86)80313-8. PMID 3782643
- [Background] Hoch DH, Batsford WP, Greenberg SM, McPherson CM, Rosenfeld LE, Marieb M, Levine JH. Double sequential external shocks for refractory ventricular fibrillation. J Am Coll Cardiol. 1994 Apr;23(5):1141-5. doi: 10.1016/0735-1097(94)90602-5. PMID 8144780
- [Background] Alaeddini J, Feng Z, Feghali G, Dufrene S, Davison NH, Abi-Samra FM. Repeated dual external direct cardioversions using two simultaneous 360-J shocks for refractory atrial fibrillation are safe and effective. Pacing Clin Electrophysiol. 2005 Jan;28(1):3-7. doi: 10.1111/j.1540-8159.2005.09155.x. PMID 15660795
- [Background] Saliba W, Juratli N, Chung MK, Niebauer MJ, Erdogan O, Trohman R, Wilkoff BL, Augostini R, Mowrey KA, Nadzam GR, Tchou PJ. Higher energy synchronized external direct current cardioversion for refractory atrial fibrillation. J Am Coll Cardiol. 1999 Dec;34(7):2031-4. doi: 10.1016/s0735-1097(99)00463-5. PMID 10588220
- [Background] Hajjar K, Berbari I, El Tawil C, Bou Chebl R, Abou Dagher G. Dual defibrillation in patients with refractory ventricular fibrillation. Am J Emerg Med. 2018 Aug;36(8):1474-1479. doi: 10.1016/j.ajem.2018.04.060. Epub 2018 Apr 30. PMID 29730094

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT03827915/Prot_SAP_ICF_000.pdf